CLINICAL TRIAL: NCT04765891
Title: Positional Release Therapy and Therapeutic Massage Reduce Muscle Trigger and Tender Points
Acronym: PRT vs TM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham Young University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ExSc PRT vs TM
Record Dates: First submitted 2021-01-12; First posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Trigger Point Pain, Myofascial
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positional Release Therapy (Experimental): Participants were randomly assigned the positional release therapy treatment group. The participants underwent the treatment.
  Interventions: Other: Positional release therapy
- Therapeutic Massage (Experimental): Participants were randomly assigned the therapeutic massage treatment group. The participants underwent the treatment.
  Interventions: Other: Therapeutic Massage

INTERVENTIONS:
Other: Positional release therapy — Positional release therapy was administered in the upper trapezius muscle. The muscle was placed in a shortened position with light pressure and held for 90 seconds per treatment location.
  Other Names: Strain Counter Strain
  Arms: Positional Release Therapy
Other: Therapeutic Massage — Participants underwent a petrissage type massage for 5 minutes at the site of the trigger point in the upper trapezius.
  Arms: Therapeutic Massage

SUMMARY:
The purpose of this study is to determine if positional release therapy (PRT) or therapeutic massage (TM) are more effective at decreasing muscle pain and tightness in the upper trapezius muscle.

DETAILED DESCRIPTION:
Introduction Myofascial pain is a common disorder affecting individuals across the general population and in specific populations, such as athletes, resulting in compromised function, performance, and productivity. It has been associated with many pain conditions including tension-type headache, spine disorder, and neck and shoulder pain. Myofascial pain characteristically results from hyperirritable nodules of muscle (trigger points or tender points) associated with pain in affected regions of the body. These areas within the muscle are subjected to continued contraction of muscle fibers due to "too much" calcium resulting in compromised oxygenation of the muscle tissue. These hyperirritable nodules often occur in fatigued muscles that are subjected to imbalanced postural positions, such as the forward head and rounded shoulders postures. It can also occur from repetitive movements commonly seen in athletics, and individuals performing manual work.

Positional release therapy (PRT) and therapeutic massage (TM) are methods used to treat trigger or tender points. Separate studies on each method have shown efficacy in reducing pain muscle tightness and improving joint mobility. PRT is a manual therapeutic technique that first locates tender points within a muscle. Once identified, the practitioner places the muscle in a passively shortened position, while applying slight pressure. TM involves the manipulation of soft tissue using techniques such as effleurage and petrissage, to restore blood flow and oxygenation of the muscle tissue.

Various methods have previously been used to find and assess severity of tender or trigger points. Among those commonly used are the pressure pain algometer with pressure pain threshold (PPT), range of motion electromyography and visual analog scales (VAS). Some studies have also utilized B-mode (two-dimensional) ultrasound imaging (US) to locate, define, trace, and quantify myofascial trigger points after palpation providing a useful means of quantification. Shear wave elastography ultrasound (SWE) has been used to calculate the elastic modulus (tissue stiffness) of muscle reliably, but has not been used quantify changes within trigger points following treatment.

Objectives The purpose of our study was to quantify the effectiveness of PRT or TM at reducing pain, trigger point tenderness, and muscle stiffness in the upper trapezius muscle by using a combination of the visual analog scale, PPT, B-mode US and SWE to assess changes within triggers points.

METHODS

Participants We recruited 60 healthy Participants, 24 males and 36 females, (age=27.1±8.8 years, wt=75.2±17.9 kg, ht= 172.8±9.7 cm) to participate in the study. Many of the participants participated on a University dance team. Participants admitted into the study were required to have upper trapezius pain, during palpation, of at least 10 mm on the 100mm visual analog scale and muscle tightness with an accompanying trigger point in their upper trapezius. Participants who had suffered an acute injury to their upper trapezius in the last 6 days, were undergoing current treatment for their upper trapezius, or were unable to lie on their stomach for an extended amount of time were removed from the study.

The study was approved by the university's Institutional Review Board before participant recruitment. All participants provided written informed consent before individual data collection began.

Instruments We used a GE LOGIC S8 ultrasound machine with the 9L soundhead to measure muscle thickness and stiffness. Muscle thickness was measured using B-mode ultrasound and SWE measured stiffness of the tissue.

In order to quantify subjective perception of pain we used PPT algometer with a .5 cm2 applicator tip along with the 100 mm visual analog scale.

Procedures During the first visit participants underwent screening for presence of inclusion and exclusion criteria as well as palpation for trigger points, following guidelines by Simons, Travell and Speicher. Each side was examined and pain produced during palpation was measured with previously published methods using the VAS. The side that was to be treated was determined by the higher VAS score. Trigger point location, found through palpation, was marked so that all measurements were taken in the same location. All baseline measurements were taken according to the methods listed below. The participants were then randomly assigned into one of two treatment groups, one being positional release therapy, the other therapeutic massage.

The same order of measurement was used for all participants since we felt that pressure from the PPT algometer could act as a treatment and influence the visual analog scale or elastography measures. Measurements were taken at rest with the participant in prone position, with their arms at their sides for all measurement series, before and after treatment.

Pain Pressure Threshold Pain pressure threshold was determined by a digital pressure algometer on the same point identified during screening. The area was measured once by pressing perpendicularly into the trigger point until the subject declared it to be painful. The peak force measured was then recorded in kg.

Ultrasound and Elastography The ultrasound machine with a 9L sound head was used to measure two different variables of muscle tension; 1) muscle thickness (B-mode) and tissue stiffness via SWE over the same spot found and marked during screening. Using B-mode on the ultrasound machine, two images aligned with the muscle fibers obtain were taken to obtain muscle thickness. Internal software was used to measure muscle thickness and the 2 images were averaged and recorded in cm. The elastography measure used a 3 cm2 box positioned over the area containing the trigger point. Nine sample circles of .5cm dimeter were set within the box side by side in rows in order to cover as much of the box as possible (shown in figure 1). (source?) Each circle registered a strain modulus reading in kPa. The average of the 9 sample circles was used to represent the stiffness of the muscle in the data analysis.

Treatment groups Therapeutic Massage Participants in the TM treatment group received a timed massage for 5 minutes by the same experienced research. A combination of effleurage and petrissage techniques were used in an organized pattern. Treatment started with effleurage (1-1.5 minutes) and proceeded to petrissage (2.5 to 3 minutes) again followed by effleurage (1 minute) over the marked area of the trigger point, but also in some surrounding areas. The pressure applied by the researcher progressed throughout the massage into the petrissage phase as tolerated by the participant and pressure was then reduced during the final effleurage phase. After the treatment was completed, the same dependent variable measurements were taken.

Positional Release Therapy Participants in the PRT group received three successive treatments or releases in the marked area. The researcher located the marked trigger point and while maintaining contact, a light pressure with the clinician's fingertip was applied creating slight dimpling of the skin and blanching of the clinician's fingernail bed. Following palpation, the researcher moved the participant's shoulder into passive abduction and scapular upward rotation and retraction until a position of comfort was achieved with no pain reported by the participant, as directed by Speicher, "Clinical Guide to Positional Release Therapy". The participant was instructed to remain completely relaxed during the 90 second treatment. After the recommended 90 seconds had passed the limb was returned to the starting position. This was repeated immediately 2 more times in tender points immediately adjacent to the first one, as recommended by Speicher. Following treatment, the same dependent variable measurements were taken.

Posttreatment measurements Each participant returned 48 hours post treatment, where dependent measurements were taken. Participants were also given an activity survey to record the number of hours they exercised between the last session and the current session to note any abnormalities or increase in normal exercise. The mark made from the first session, over the examined trigger point, was still visible at the second visit for all participants and was used to determine the location for performing dependent measurements.

Statistical Analysis A mixed-models analysis of variance was performed for each of the dependent variables (VAS, US, elastography, and PPT). The covariates considered in the analysis were the participants' sex, side of treatment, height, weight, and age. A step-wise regression was used to determine significant covariates for each of the dependent variables. Following the step-wise regression the primary variables of interest, treatment and time of measurement were added along with their interaction for each of the dependent variables. Post hoc t-tests were used to evaluate differences in the measurements. All analyses were performed using SAS, version 9.4 and alpha was set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* dancers at the university
* Subjects experiencing upper trapezius pain and muscle tightness, with associated tender or trigger points
* Need to be able to lie on stomach for at least 30 minutes
* Not be currently receiving treatment from the Dance Athletic Training Room on their trapezius.

Exclusion Criteria:

* Pregnant
* Unable to lie on stomach for 30 minutes
* Currently be receiving treatment on their upper trapezius muscle.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2018-02-09 (Actual); Study Completion 2018-02-09 (Actual)

PRIMARY OUTCOMES:
Pain perception | 72 hours
  Rating of perceived pain as measured by the visual analog scale (VAS) on a scale of 0 to 100. With 100 being the highest pain score.
Pain Pressure Threshold (PPT) | 72 hours
  Pressure was measured by an algometer on a continuous scale. A higher score would indicate an individual tolerating more pressure.
Tissue Stiffness | 72 Hours
  Tissue stiffness was measured using Shear Wave Elastography on a scale of 0 150, with larger numbers indicating a higher tissue stiffness.
Muscle Thickness | 72 hours
  B-Mode Ultrasound was used to measure the resting thickness of the trapezius. muscle

CONTACTS AND LOCATIONS:
Overall Officials: Aaron W Johnson, PhD, Principal Investigator — Associate Professor
Locations (1):
- Brigham Young University, Provo, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
If data is requested through e-mail by another investigator or institution, and approved by the institutional review board then data will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will become available upon e-mail request. This will be for at least 3 years.
Access Criteria: E-mail to principal investigator from validated researchers.

REFERENCES:
- [Background] Aboodarda SJ, Spence AJ, Button DC. Pain pressure threshold of a muscle tender spot increases following local and non-local rolling massage. BMC Musculoskelet Disord. 2015 Sep 28;16:265. doi: 10.1186/s12891-015-0729-5. PMID 26416265
- [Background] Borg-Stein J, Simons DG. Focused review: myofascial pain. Arch Phys Med Rehabil. 2002 Mar;83(3 Suppl 1):S40-7, S48-9. doi: 10.1053/apmr.2002.32155. PMID 11973695
- [Background] Buttagat V, Eungpinichpong W, Chatchawan U, Arayawichanon P. Therapeutic effects of traditional Thai massage on pain, muscle tension and anxiety in patients with scapulocostal syndrome: a randomized single-blinded pilot study. J Bodyw Mov Ther. 2012 Jan;16(1):57-63. doi: 10.1016/j.jbmt.2011.04.005. Epub 2011 Jun 22. PMID 22196428
- [Background] Cojocaru MC, Cojocaru IM, Voiculescu VM, Cojan-Carlea NA, Dumitru VL, Berteanu M. Trigger points--ultrasound and thermal findings. J Med Life. 2015 Jul-Sep;8(3):315-8. PMID 26351532
- [Background] D'Ambrogio KJ, Roth GB 1997 Positional Release Therapy. Mosby.
- [Background] Dommerholt J, Bron C, Franssen J 2006 Myofascial trigger points: an evidence-informed review. Journal of Manual & Manipulative Therapy 14, 203-221.
- [Background] Draper D 2015 The Deep Muscle Stimulator's Effects on Tissue Stiffness in Trigger-Point Therapy. Athletic Therapy Today 10, 52-53.
- [Background] Ghanbari A, Rahimijaberi A, Mohamadi M, Abbasi L, Sarvestani FK. The effect of trigger point management by positional release therapy on tension type headache. NeuroRehabilitation. 2012;30(4):333-9. doi: 10.3233/NRE-2012-0764. PMID 22672949
- [Background] Jafri MS. Mechanisms of Myofascial Pain. Int Sch Res Notices. 2014;2014:523924. doi: 10.1155/2014/523924. PMID 25574501
- [Background] JG T, SH R 1983 Myofascial pain and dysfunction: the trigger point manual. Williams & Wilkins, Baltimore MD.
- [Background] Kelencz CA, Tarini VA, Amorim CF. Trapezius upper portion trigger points treatment purpose in positional release therapy with electromyographic analysis. N Am J Med Sci. 2011 Oct;3(10):451-5. doi: 10.4297/najms.2011.3451. PMID 22363082
- [Background] Knight KL, Draper DO 2013 Therapeutic Modalities: The Art and Science. Lippincott Williams & Wilkins, Baltimore, MD.
- [Background] Kumbhare DA, Elzibak AH, Noseworthy MD. Assessment of Myofascial Trigger Points Using Ultrasound. Am J Phys Med Rehabil. 2016 Jan;95(1):72-80. doi: 10.1097/PHM.0000000000000376. PMID 26334421
- [Background] Mohammadi Kojidi M, Okhovatian F, Rahimi A, Baghban AA, Azimi H. The influence of Positional Release Therapy on the myofascial trigger points of the upper trapezius muscle in computer users. J Bodyw Mov Ther. 2016 Oct;20(4):767-773. doi: 10.1016/j.jbmt.2016.04.006. Epub 2016 Apr 7. PMID 27814857
- [Background] Muller CE, Aranha MF, Gaviao MB. Two-dimensional ultrasound and ultrasound elastography imaging of trigger points in women with myofascial pain syndrome treated by acupuncture and electroacupuncture: a double-blinded randomized controlled pilot study. Ultrason Imaging. 2015 Apr;37(2):152-67. doi: 10.1177/0161734614546571. Epub 2014 Aug 12. PMID 25116293
- [Background] Nagrale AV, Glynn P, Joshi A, Ramteke G. The efficacy of an integrated neuromuscular inhibition technique on upper trapezius trigger points in subjects with non-specific neck pain: a randomized controlled trial. J Man Manip Ther. 2010 Mar;18(1):37-43. doi: 10.1179/106698110X12595770849605. PMID 21655422
- [Background] Myofascial trigger points, a possible explanation. Pain. 1981 Feb;10(1):106-109. doi: 10.1016/0304-3959(81)90053-1. No abstract available. PMID 7232007
- [Background] Sweety CC, Vinod KB, Kumar NS, Ayyappan V 2014 Effect of Positional Release Technique in Subjects with Subacute Trapezitis. Int J Physiother 1, 91-99.
- [Background] Tessier DG 2005 Sports massage: An overview. International Journal of Athletic Therapy and Training 10, 67-69.
- [Background] Wong CK. Strain counterstrain: current concepts and clinical evidence. Man Ther. 2012 Feb;17(1):2-8. doi: 10.1016/j.math.2011.10.001. Epub 2011 Oct 24. PMID 22030379

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-08-04): https://cdn.clinicaltrials.gov/large-docs/91/NCT04765891/Prot_SAP_000.pdf
  • Informed Consent Form (2017-07-07): https://cdn.clinicaltrials.gov/large-docs/91/NCT04765891/ICF_001.pdf